CLINICAL TRIAL: NCT02039011
Title: Proof of Concept Study to Evaluate Single and Chronic Dosing Effects of Ultra-long Acting Bronchodilator Therapy on Mannitol Challenge in Asthmatic Patients Taking Inhaled Corticosteroids
Brief Title: Ultra-long Acting Bronchodilator Therapy in Asthmatics
Acronym: MAN02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Tenovus Scotland (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor of Allergy and Pulmonology, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012RC15
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Long acting beta-agonists; Long acting muscarinic antagonists; Mannitol challenge
MeSH Terms: conditions — Asthma | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol (Active Comparator)
  Interventions: Drug: Indacaterol
- Indacaterol & tiotropium (Experimental)
  Interventions: Drug: Indacaterol and tiotropium

INTERVENTIONS:
Drug: Indacaterol — Participants receive indacaterol for 2 to 4 weeks. Participants then enter a washout period and after the washout period receive the alternative treatment arm.
  Arms: Indacaterol
Drug: Indacaterol and tiotropium — Participants receive indacaterol and tiotropium for 2 to 4 weeks. Participants then enter a washout period and after the washout period receive the alternative treatment arm.
  Arms: Indacaterol & tiotropium

SUMMARY:
Asthma is a common condition which produces a significant workload for general practice, hospital outpatient clinics and inpatient admissions. Asthma is caused by inflammation of the airways which irritates the muscles around the airways causing them to constrict. The mainstay of asthma treatment is inhaled steroids. If the patients' symptoms are still not adequately controlled, then a long-acting beta agonist (LABA) inhaler which relaxes the muscles in the airways and opens it up is frequently added to the inhaled steroids. Despite this, a substantial proportion of asthmatic patients still do not achieve adequate control of their symptoms. Recent studies have shown when an alternative inhaler called a long-acting muscarinic antagonist (LAMA) is added to a LABA - it reduced the number of asthma exacerbations (flare-ups) and improved airway narrowing.

The mannitol challenge is a test of airway 'twitchiness', an important feature of asthma. There have been no previous studies assessing the combined effects LABA and LAMA inhalers on mannitol challenge. The mannitol challenge is particularly relevant as it mimics stimuli encountered in real life which provoke an asthma attack.

The investigators propose to directly compare indacaterol, a new once-daily LABA with indacaterol plus tiotropium, a once-daily LAMA, as add-on treatment to inhaled steroids in persistent asthmatics using the mannitol challenge. The investigators hope that this study will help us understand how the combination of a LABA and LAMA might help protect against flare-ups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged at least 16 years with persistent asthma and on inhaled corticosteroids (at least 400 micrograms of beclomethasone dipropionate or the equivalent
* FEV1 > 50 % predicted
* Mannitol PD15 < 635 mg
* Ability to give informed consent
* Agreement for their general practitioner to be made aware of study participation and to receive feedback as relevant to the participant's well being

Exclusion Criteria:

* Other respiratory diseases such as chronic obstructive pulmonary disease, bronchiectasis or allergic bronchopulmonary aspergillosis
* An asthma exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 3 months of the study commencement
* Any clinically significant medical condition that may endanger the health or safety of the participant
* Smoking within one year or >10 pack year history
* Participation in another trial within 30 days before the commencement of the study
* Pregnancy or lactation
* Unable to comply with the procedures of the protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in provocation dose of mannitol causing 15% drop in forced expiratory volume in 1 second (PD15) between single and chronic dosing of ultra-long acting bronchodilator therapy | 2 to 4 weeks

SECONDARY OUTCOMES:
Mannitol Response-dose Ratio (RDR) | 2 to 4 weeks
Salbutamol recovery time following mannitol challenge | 2 to 4 weeks
Domiciliary peak expiratory flow (PEF) | 2 to 4 weeks
Trough forced expiratory volume in 1 second (FEV1) | 2 to 4 weeks
Exhaled nitric oxide (FeNO) | 2 to 4 weeks
Trough impulse oscillometry (IOS) | 2 to 4 weeks
Asthma Control Questionnaire (ACQ) | 2 to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, Principal Investigator — University of Dundee; Arvind Deva Manoharan, MBChB, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Result] Jabbal S, Manoharan A, Lipworth BJ. Bronchoprotective tolerance with indacaterol is not modified by concomitant tiotropium in persistent asthma. Clin Exp Allergy. 2017 Oct;47(10):1239-1245. doi: 10.1111/cea.12972. Epub 2017 Aug 1. PMID 28665534